CLINICAL TRIAL: NCT06526182
Title: A Phase 3, 2-Part, Open-Label and Double-Blind, Randomised Study to Evaluate the Effectiveness and Safety of Lebrikizumab Treatment in Adults and Adolescents With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study of Lebrikizumab Treatment in Adults and Adolescents With Moderate-to-Severe Atopic Dermatitis
Acronym: ADhope 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M-17923-34; 2023-508235-31 (EudraCT Number)
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Dermatitis, Atopic; Eczema
Keywords: Dermatitis; Skin Diseases; Skin Diseases, Eczematous; Moderate-to-severe atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Skin Diseases; Skin Diseases, Eczematous | interventions — lebrikizumab

STUDY DESIGN:
Intervention Model Description: Part 1 and Part 2 (Run-In Period): Open label; Part 2: Randomized and Double-Blind.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Part 1: Open label (Lebrikizumab) (Experimental): Participants with moderate-to-severe AD will receive loading doses of lebrikizumab 500 mg SC injection (2 injections) at Day 1 and Week 2 followed by 250 mg (1 injection) every 2 weeks (Q2W) after Week 4 to Week 16 followed by 250 mg (1 injection) every 4 weeks (Q4W) after Week 16 to Week 24.
  Interventions: Biological: Lebrikizumab
- Part 2: Open label Run-In Period (Lebrikizumab) (Experimental): Participants who respond to lebrikizumab treatment at Week 24 of Part 1 will continue treatment in Part 2, which includes an 8-week open-label Run-In Period to confirm sustained clinical response. During this period, they will receive lebrikizumab 250 mg SC injection (1 injection) Q4W starting from the Week 24 visit of Part 1.
  Interventions: Biological: Lebrikizumab
- Part 2: Double-Blind (Lebrikizumab) (Experimental): At the end of the Run-In Period, participants who demonstrate sustained clinical response will continue treatment in the double-blind period. They will either receive lebrikizumab 250 mg SC injection (1 injection) Q4W or switch to lebrikizumab 500 mg SC injection (2 injections) Q12W for 36 weeks.
  Interventions: Biological: Lebrikizumab
- Part 2: Double-Blind (Placebo) (Placebo Comparator): At the end of the Run-In Period, participants who demonstrate sustained clinical response will continue treatment in the double-blind period. They will either receive lebrikizumab matching placebo 250 mg SC injection (1 injection) Q4W or switch to lebrikizumab matching placebo 500 mg SC injection (2 injections) Q12W for 36 weeks.
  Interventions: Other: Placebo
- Part 2: Open label Escape Arm (Lebrikizumab) (Experimental): Participants who do not maintain at least a 50% reduction in EASI from baseline (EASI 50) during Double-Blind Period will enter an Escape Arm, in which participants are treated with open label lebrikizumab 250 mg SC injection Q4W. Study drug treatment will be discontinued in participants entering the Escape Arm who do not maintain an EASI 50 response.
  Interventions: Biological: Lebrikizumab

INTERVENTIONS:
Biological: Lebrikizumab — Lebrikizumab solution for injection administered subcutaneously.
  Arms: Part 1: Open label (Lebrikizumab); Part 2: Double-Blind (Lebrikizumab); Part 2: Open label Escape Arm (Lebrikizumab); Part 2: Open label Run-In Period (Lebrikizumab)
Other: Placebo — Lebrikizumab Matching placebo solution for injection administered subcutaneously.
  Arms: Part 2: Double-Blind (Placebo)

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of 24 weeks of lebrikizumab in improving disease severity, signs, and symptoms in adults and adolescents with moderate-to-severe AD in Part 1 and to describe how similar is the current maintenance dosing regimen of lebrikizumab 250 mg every 4 weeks (Q4W) to the new proposed; lebrikizumab 500 mg every 12 weeks (Q12W), in terms of efficacy, safety, PK, ADA and blood biomarkers.

DETAILED DESCRIPTION:
This study consists of two parts. Part 1 is a single-arm, open-label design, where participants will receive lebrikizumab subcutaneous (SC) injections up to Week 24. Part 2 is a randomized, double-blind design, in which participants who achieve clinical response in Part 1 will continue receiving lebrikizumab treatment across two periods: a Run-in period and a Double-blind period. Participants who do not maintain at least a 50% reduction in Eczema Area and Severity Index (EASI) from baseline during Double-Blind Period will enter an Escape Arm.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

1. Adults and adolescents (aged greater than or equal to [>=] 12 to less than [<] 18 at the time of informed consent form [ICF]/informed assent form [IAF] signature and weighing 40 >= kilograms [kg]) who are candidates for systemic AD therapy.
2. Chronic AD (according to Hanifin and Rajka Criteria (Hanifin 1980)) that has been present for >= 1 year before the screening visit.
3. EASI score >= 12 at the Day 1/Baseline Visit.
4. IGA score >= 3 (moderate) (scale of 0 [clear] to 4 [severe]) at the Day 1/Baseline visit.
5. >= 10% BSA of AD involvement at the Day 1/Baseline visit.
6. History of inadequate response to treatment with topical medications; or determination that topical treatments are otherwise medically inadvisable.
7. Completed electronic diary (eDiary) entries for pruritus and sleep-loss for a minimum of 4 of 7 days before Day 1/Baseline.
8. Willing and able to comply with all clinic visits and study-related procedures and questionnaires.
9. For women of childbearing potential: agree to remain abstinent (refrain from heterosexual intercourse) or to use a highly effective contraceptive method during the treatment period and for at least 4 weeks or 1 menstrual period after the last dose of lebrikizumab.
10. Participant must provide signed ICF. Adolescent participants must also provide separate informed assent to enroll in the study and sign and date either a separate IAF or the ICF signed by the parent/legal guardian (as appropriate based on local regulations and requirements).

    Part 2:
11. Demonstrate clinical response to treatment at Week 24 of Part 1, defined as achieving EASI 75 or IGA 0/1 without the use of high-potency TCS within the prior 4 weeks or systemic corticosteroids at any time post baseline.

Exclusion Criteria:

1. Prior treatment at any time with tralokinumab, lebrikizumab, or an oral JAK inhibitor.
2. Intention to use any concomitant medication or therapy that is not permitted by this protocol or failure to undergo the required washout period for a particular prohibited medication.
3. History of anaphylaxis as defined by the Sampson criteria (Sampson 2006).
4. Uncontrolled chronic disease that might require bursts of oral corticosteroids, eg, comorbid severe uncontrolled asthma (defined by an Asthma Control Questionnaire-5 score >= 1.5 or a history of >= 2 asthma exacerbations within the last 12 months requiring systemic [oral and/or parenteral] corticosteroid treatment or hospitalisation for >24 hours).
5. Occurrence of the following types of infection within 3 months before or during screening or development of these infections before Day 1/Baseline:

   1. Serious (requiring hospitalisation, and/or IV or equivalent oral antibiotic treatment, as per the Investigator's opinion);
   2. Opportunistic (as defined by Winthrop et al. (Winthrop 2015))
   3. Chronic (duration of symptoms, signs, and/or treatment of 6 weeks or longer);
   4. Recurring (including, but not limited to herpes simplex, herpes zoster, recurring cellulitis, chronic osteomyelitis).
6. Known current or chronic infection with any hepatitis virus.
7. Known liver cirrhosis and/or chronic hepatitis of any aetiology.
8. Known active endoparasitic infection or at high risk of these infections.
9. Known or suspected history of immunosuppression, including history of invasive opportunistic infections (e.g., tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, and aspergillosis) despite infection resolution: or unusually frequent, recurrent, or prolonged infections, per the Investigator's judgement.
10. History of human immunodeficiency virus (HIV) infection or known positive HIV serology.
11. Any clinically significant laboratory test results from the chemistry or haematology tests obtained at the Screening visit that would jeopardise the participants participation in the study, per the Investigator's judgement.
12. Presence of skin comorbidities that may interfere with study assessments.
13. History of malignancy, including mycosis fungoides, within 5 years before the Screening visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved nonmetastatic squamous or basal cell carcinoma of the skin with no evidence of recurrence in the past 12 weeks.
14. Severe concomitant illness(es) that in the Investigator's judgement would adversely affect the participation in the study. Any other medical or psychological condition that in the opinion of the Investigator may suggest a new and/or insufficiently understood disease, may present an unreasonable risk to the study participant because of his/her participation in this clinical trial, may make participation unreliable, or may interfere with study assessments.
15. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.
16. Any known hypersensitivity or allergic response to lebrikizumab or any component of the investigational medicinal product (IMP).
17. For the scratch sensor substudy only: a history of allergic response to skin adhesives, active skin or systemic infection, active AD on the back of the hand, or a pre-existing sleep disorder, including insomnia, obstructive sleep apnea, or restless leg syndrome, or currently taking prescription sleep medications.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Part 1: Percentage of Participants Achieving Eczema Area and Severity Index (EASI) Score Less than or Equal to (<=) 7 at Week 24 | At Week 24
  The EASI is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and or extensive disease. The severity of erythema, induration/papulation, excoriation, and lichenification will be assessed by the Investigator or trained designee on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. In addition, the extent of AD involvement in each of the 4 body areas will be assessed as a percentage by body area of head/neck, trunk, upper limbs, and lower limbs, and converted to a score of 0 (0%), 1 (0 to 9%), 2 (10 to 29%), 3 (30 to 49%), 4 (50 to 69%), 5 (70 to 89%) and 6 (90 to 100%).
Part 2: Percentage of Participants Achieving EASI 75 at Week 36 | At Week 36
  The EASI is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and or extensive disease. EASI 75 is defined as 75% reduction from baseline in the EASI score.
Part 2: Percentage of Participants with an IGA Score of 0 or 1 and a Reduction >=2 Points | From Baseline (Part 1) up to Week 36
  The IGA is an instrument used to globally rate the severity of the participant's AD. It is based on a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate) and 4 (severe), and a score is selected using descriptors that best describe the overall appearance of the lesions at a given time point. The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting (minimal, palpable induration and significant induration).

SECONDARY OUTCOMES:
Part 1: Time to Achieve an EASI Score <= 7 | Baseline up to Week 24
  The EASI is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and or extensive disease.
Part 1: Percentage of Participants Achieving EASI <=5, and EASI <=3 at Week 24 | At Week 24
  The EASI is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and or extensive disease. The severity of erythema, induration/papulation, excoriation, and lichenification will be assessed by the Investigator or trained designee on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. In addition, the extent of AD involvement in each of the 4 body areas will be assessed as a percentage by body area of head/neck, trunk, upper limbs, and lower limbs, and converted to a score of 0 (0%), 1 (0 to 9%), 2 (10 to 29%), 3 (30 to 49%), 4 (50 to 69%), 5 (70 to 89%) and 6 (90 to 100%).
Part 1: Percentage of Participants Achieving EASI 75 and EASI 90 at Week 24 | At Week 24
  The EASI is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and or extensive disease. EASI 75 is defined as 75% reduction from baseline in the EASI score. EASI 90 is defined as 90% reduction from baseline in the EASI score.
Part 1: Percentage of Participants with an Investigator Global Assessment (IGA) Score of 0 or 1 and a Reduction Greater Than or Equal to (>=2) Points at Week 24 | At Week 24
  The IGA is an instrument used to globally rate the severity of the participant's AD. It is based on a 5-point scale ranging from 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate) and 4 (severe), and a score is selected using descriptors that best describe the overall appearance of the lesions at a given time point. The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting (minimal, palpable induration and significant induration).
Part 1: Percentage of Participants Achieving Scoring Atopic Dermatitis (SCORAD) 75, and SCORAD 90 at Week 24 | At Week 24
  The SCORAD is a validated measure of the extent and severity of atopic dermatitis lesions, along with subjective symptoms. The score ranges from 0 to 103, with higher values indicating a more extensive and/or severe condition. SCORAD 75 is defined as 75% reduction in SCORAD from baseline. SCORAD 90 is defined as 90% reduction in SCORAD from baseline.
Part 1: Percentage Change From Baseline in Modified Total Lesion Symptom Score (mTLSS) at Week 24 | At Week 24
  mTLSS combines an evaluation of hand eczema lesions severity including 6 key signs (erythema, desquamation, lichenification/hyperkeratosis, vesiculae, oedema, fissures) and the intensity of pruritus and pain. The seven features of AD of the hand (erythema, scaling, lichenification/hyperkeratosis, vesiculation, oedema, fissures, pruritus/pain) form the composite scale of mTLSS' strength and each one of them scores from 0 (mild) to 3 (severe). The scores is summed, extending from a base estimation of 0 (no signs or symptoms) to the most extreme of 21 (more serious disease).
Part 1: Percentage of Participants with Pruritus Numerical Rating Scale (NRS) >=4 at Baseline Achieving >=4-Point Improvement in Pruritus NRS | Baseline up to Week 24
  The Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours, with 0 indicating "No itch," and 10 indicating "Worst itch imaginable.
Part 1: Percentage of Participants Achieving Dermatology Life Quality Index (DLQI) 0-1 at Week 24 | At Week 24
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicates 0-1 (no effect on patient's life), 2-5 (small effect on patient's life), 6-10 (moderate effect on patient's life), 11-20 (very large effect on patient's life), 21-30 (extremely large effect on patient's life)
Part 1: Percentage of Participants Achieving Children Dermatology Life Quality Index (cDLQI) 0-1 at Week 24 | At Week 24
  cDLQI is validated from adolescents younger than age of 16 years, which is based on a set of 10 questions different from those of the DLQI. The answers to the questions are generally scored on a 4-point scale from 0=not at all or question unanswered, 1=only a little, 2=quite a lot, 3=very much. cDLQI is calculated by summing the score of each question resulting in 0 to 30. Higher the score, the more impairment of the child's life is experienced.
Part 1: Percentage of Participants with DLQI >=4 at Baseline Achieving >=4-Point Improvement in DLQI | Baseline up to Week 24
  DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. High score is indicative of a poor QoL.
Part 1: Percentage of Participants with cDLQI >=6 at Baseline Achieving >=6-Point Improvement in cDLQI | Baseline up to Week 24
  cDLQI is validated from adolescents younger than age of 16 years, which is based on a set of 10 questions different from those of the DLQI. The answers to the questions are generally scored on a 4-point scale from 0=not at all or question unanswered, 1=only a little, 2=quite a lot, 3=very much. cDLQI is calculated by summing the score of each question resulting in 0 to 30. Higher the score, the more impairment of the child's life is experienced.
Part 1: Percentage of Participants with a Sleep-Loss Scale of >=2 Points at Baseline Achieving >= 2 Point Improvement at Week 24 | At Week 24
  Sleep loss will be assessed by all participants using a patient-related outcome (PRO) instrument. Participants (and if applicable, with help of parents/caregiver if required) will rate their sleep on a 5-point Likert scale (with scores ranging from 0 [not at all] to 4 [unable to sleep at all]). Assessments will be recorded by the participant using an eDiary. The baseline Sleep-Loss Scale score will be determined based on the average of daily Sleep-Loss Scale scores during the 7 days immediately before the Day 1 or Baseline visit.
Part 1: Percentage of Participants with Patient-Oriented Eczema Measure (POEM) >=4 at Baseline Achieving >=4-Point Improvement in POEM | Baseline up to Week 24
  The POEM is a 7-item, validated questionnaire completed by the participant (and, if applicable, with help of parents/caregiver if required) to assess disease symptoms. Participants are asked to respond to questions on skin dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping. All answers carry equal weight, with a total possible score ranging from 0 to 28 (answers scored as: No days = 0; 1-2 days = 1; 3-4 days = 2; 5-6 days = 3; every day = 4. A high score is indicative of a poor quality of life. POEM responses will be captured weekly using an eDiary.
Part 1: Percentage of Participants with Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Related AEs, AEs Leading to Study Treatment Discontinuation, and Adverse Events of Special Interest (AESIs) | Baseline up Week 24
  An AE is defined as any untoward medical occurrence in a clinical trial participant, regardless of the administration of the IMP and its causal relationship to it. An AE can therefore be any unfavourable/unintended medical occurrence during the participation in the trial, including deterioration of a pre-existing medical condition, an abnormal value in a laboratory assessment, ECG abnormality, or an abnormal finding in the physical examination. An SAE is an AE, which falls into any of the following categories: death, is life-threatening, requires in-patient hospitalisation or prolongs existing hospitalisation, persistent or significant disability or incapacity, congenital anomaly or birth defect, or any other medically important event that may jeopardise the participant or may require intervention to prevent one of the other above outcomes. The following treatment-emergent AEs are being designated as AESIs: conjunctivitis, herpes simplex or zoster infection and parasitic infections.
Part 2: Percentage of Participants Achieving EASI Scores <=7, and <=3 at Week 36 | At Week 36
  The EASI is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and or extensive disease. The severity of erythema, induration/papulation, excoriation, and lichenification will be assessed by the Investigator or trained designee on a scale of 0 (absent) to 3 (severe) for each of the 4 body areas: head/neck, trunk, upper limbs, and lower limbs, with half points allowed. In addition, the extent of AD involvement in each of the 4 body areas will be assessed as a percentage by body area of head/neck, trunk, upper limbs, and lower limbs, and converted to a score of 0 (0%), 1 (0 to 9%), 2 (10 to 29%), 3 (30 to 49%), 4 (50 to 69%), 5 (70 to 89%) and 6 (90 to 100%).
Part 2: Percentage of Participants Achieving EASI 90 at Week 36 | At Week 36
  The EASI is used to assess the severity and extent of AD; it is a composite index with scores ranging from 0 to 72, with higher values indicating more severe and or extensive disease. EASI 90 is defined as 90% reduction from baseline in the EASI score.
Part 2: Percentage of Participants with Pruritus NRS >=4 at Baseline (Part 1) Achieving >=4-Point Improvement in Pruritus NRS at Week 36 | At Week 36
  The Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours, with 0 indicating "No itch," and 10 indicating "Worst itch imaginable.
Part 2: Percentage of Participants with Pruritus NRS 0 or 1 at Week 36 | At Week 36
  The Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours, with 0 indicating "No itch," and 10 indicating "Worst itch imaginable.
Part 2: Percentage of Participants Achieving DLQI 0-1 at Week 36 | At Week 36
  The DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. A high score is indicative of a poor QoL. DLQI scores indicates 0-1 (no effect on patient's life), 2-5 (small effect on patient's life), 6-10 (moderate effect on patient's life), 11-20 (very large effect on patient's life), 21-30 (extremely large effect on patient's life).
Part 2: Percentage of Participants Achieving cDLQI 0-1 at Week 36 | At Week 36
  cDLQI is validated from adolescents younger than age of 16 years, which is based on a set of 10 questions different from those of the DLQI. The answers to the questions are generally scored on a 4-point scale from 0=not at all or question unanswered, 1=only a little, 2=quite a lot, 3=very much. cDLQI is calculated by summing the score of each question resulting in 0 to 30. Higher the score, the more impairment of the child's life is experienced.
Part 2: Percentage of Participants with DLQI >=4 at Baseline (Part 1) Achieving >=4-Point Improvement in DLQI at Week 36 | At Week 36
  DLQI is a 10-item validated questionnaire completed by the participant or caregiver used to assess the impact of skin disease on the participant's QoL during the previous week. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment. Each question is scored from 0=not at all, 1=a little, 2=a lot, and 3=very much, giving a total score ranging from 0 to 30. High score is indicative of a poor QoL.
Part 2: Percentage of Participants with cDLQI >=6 at Baseline (Part 1) Achieving >=6-Point Improvement in cDLQI at Week 36 | At Week 36
  cDLQI is validated from adolescents younger than age of 16 years, which is based on a set of 10 questions different from those of the DLQI. The answers to the questions are generally scored on a 4-point scale from 0=not at all or question unanswered, 1=only a little, 2=quite a lot, 3=very much. cDLQI is calculated by summing the score of each question resulting in 0 to 30. Higher the score, the more impairment of the child's life is experienced.
Part 2: Percentage of Participants with a Sleep-Loss Scale of >=2 Points at Baseline (Part 1) Achieving >= 2 Point Improvement at Week 36 | At Week 36
  Sleep loss will be assessed by all participants using a PRO instrument. Participants (and if applicable, with help of parents/caregiver if required) will rate their sleep on a 5-point Likert scale (with scores ranging from 0 [not at all] to 4 [unable to sleep at all]). Assessments will be recorded by the participant using an eDiary. The baseline Sleep-Loss Scale score will be determined based on the average of daily Sleep-Loss Scale scores during the 7 days immediately before the Day 1 or Baseline visit.
Part 2: Percentage of Participants with POEM >=4 at Baseline (Part 1) Achieving >=4-Point Improvement in POEM at Week 36 | At Week 36
  The POEM is a 7-item, validated questionnaire completed by the participant (and, if applicable, with help of parents/caregiver if required) to assess disease symptoms. Participants are asked to respond to questions on skin dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping. All answers carry equal weight, with a total possible score ranging from 0 to 28 (answers scored as: No days = 0; 1-2 days = 1; 3-4 days = 2; 5-6 days = 3; every day = 4. A high score is indicative of a poor quality of life. POEM responses will be captured weekly using an eDiary.
Part 2: Percentage of Participants with TEAEs, SAEs, Related AEs, AEs Leading to Study Treatment Discontinuation, and AESIs | From Week 24 up to Week 68
  An AE is defined as any untoward medical occurrence in a clinical trial participant, regardless of the administration of the IMP and its causal relationship to it. An AE can therefore be any unfavourable/unintended medical occurrence during the participation in the trial, including deterioration of a pre-existing medical condition, an abnormal value in a laboratory assessment, ECG abnormality, or an abnormal finding in the physical examination. An SAE is an AE, which falls into any of the following categories: death, is life-threatening, requires in-patient hospitalisation or prolongs existing hospitalisation, persistent or significant disability or incapacity, congenital anomaly or birth defect, or any other medically important event that may jeopardise the participant or may require intervention to prevent one of the other above outcomes. The following treatment-emergent AEs are being designated as AESIs: conjunctivitis, herpes simplex or zoster infection and parasitic infections.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Almirall, S.A.
Locations (4):
- Spain (4):
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital del Mar - Parc de Salut Mar, Barcelona
  - Hospital Universitario Clínico San Cecilio, Granada
  - Consorci Hospital General Universitari de València, Valencia

IPD SHARING:
Plan to Share IPD: No